CLINICAL TRIAL: NCT02969343
Title: Patient Safety Learning Laboratory: Making Acute Care More Patient-Centered
Acronym: PSLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Principal Investigator, David W. Bates, MD, MSc, Senior Vice President and Chief Innovation Officer, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5P30HS023535 (AHRQ)
Record Dates: First submitted 2016-10-24; First posted 2016-11-21 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Central Line-Associated Bloodstream Infection (CLABSI); Venous Thromboembolism; Patient Fall; Catheter-Associated Infection; Severe Hypoglycemia; Opioid-Related Severe Adverse Drug Event; Hospital Acquired Pressure Ulcer; Adverse Drug Event; Severe Hospital Acquired Delerium; Rapid Response Related to Arrhythmia
MeSH Terms: conditions — Venous Thromboembolism; Catheter-Related Infections; Hypoglycemia; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients and providers on hospital care units where the PSLL patient safety health information technology tools are implemented, during the interventional phase of a stepped wedge randomized trial design.
  Interventions: Behavioral: Patient Safety health information technology
- Usual Care (No Intervention): Patients on hospital care units where the PSLL patient safety health information technology tools have been implemented or are to be implemented, but are not during the usual care phase of a stepped wedge randomized trial design.

INTERVENTIONS:
Behavioral: Patient Safety health information technology — Patient safety technology toolkits on hospital care units
  Arms: Intervention

SUMMARY:
The Brigham and Women's Hospital (BWH) Patient Safety Learning Laboratory (PSLL) focuses on developing health information technology (HIT) tools to engage patients, family, and professional care team members in reliable identification, assessment, and reduction of patient safety threats in real-time, before they manifest in actual harm.

DETAILED DESCRIPTION:
The Brigham and Women's Hospital (BWH) Patient Safety Learning Laboratory (PSLL) will develop systems approaches to integrating health information technology (HIT), stakeholder engagement mechanisms, and process design/engineering methods focused on patient safety, development and enhancement of tools, health care system interventions, and translation into practice. The three technological toolkits to be developed as part of the Patient Safety Learning Laboratory (PSLL) are:1) Patient-centered Fall Prevention Toolkit which aims to engage patients and their family caregivers in the design of HIT tools to prevent patient falls and related injuries during an acute hospitalization; 2) Patient Safety Checklist Tool to improve patient safety and quality outcomes, provider efficiency, and team communication; and 3) MySafeCare Patient Safety Reporting System which aims to iteratively develop and evaluate the impact of a patient safety reporting system on patient safety and fosters a health system focused on collaborative learning. The Brigham and Women's Patient Safety Learning Laboratory (BWH PSLL) will establish a vibrant learning ecosystem of health services, informatics, and systems engineering researchers, collaborating with patients and family for evolving and applying these approaches to adverse event prevention in hospitalized patients. In addition, a Systems Engineering, Usability, and Integration (SEUI) Core will leverage health systems engineering approaches to develop and provide a system-wide methodology to aid in the successful implementation and improvement of Health Information Technology (HIT) tools and a model known as the Patient SatisfActive® will be developed, tested, and refined to create a culture of patient- and family-centered care.

ELIGIBILITY:
Inclusion Criteria:

* patients 18-99 years of age

Exclusion Criteria:

* patients under age 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21000 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes: Proportion of hospitalizations with any adverse event | up to 21 months
  Hospitalizations with the presence of any of the following: Patient Falls with Injury, Severe Hypoglycemia, Inpatient or post hospitalization venous thromboembolism, catheter associated urinary tract infection (CAUTI), Central Line Associated Blood Stream Infection (CLABSI), Opioid related severe adverse drug event, hospital acquired pressure ulcer, severe hospital acquired delirium, rapid response related to arrhythmia

SECONDARY OUTCOMES:
Clinical Inertia: When Red flag, % changed to yellow or green during hospitalization | up to 21 months
  monitoring time for flags to change within patient safety information technology tools
Clinical Inertia:When Red flag, % changed to green during hospitalization | up to 21 months
  monitoring time for flags to change within patient safety information technology tools
Clinical Inertia: Mean time to resolution of red flags (to green or yellow), days | up to 21 months
  monitoring time for flags to change within patient safety information technology tools
Clinical Inertia:Mean time to resolution of red flags (to green), days | up to 21 months
  monitoring time for flags to change within patient safety information technology tools
Patient Falls/ Mobility: % patient days of patients at fall risk due to a gait disturbance on sedatives | up to 21 months
  Processes of care: % patient days of patients at fall risk due to a gait disturbance on sedatives
Patient Falls/ Mobility:% pt-days of patients at fall risk due to a gait disturbance without Physical Therapy consult order | up to 21 months
  Processes of care: % patient-days of patients at fall risk due to a gait disturbance without Physical Therapy consult order
Code Status: % patient-days on study unit with unconfirmed code status | up to 21 months
  Processes of care: % patient-days on study unit with unconfirmed code status
Glucose Control: % patients with diabetes or hyperglycemia with order for basal insulin | up to 21 months
  Processes of care: % patients with diabetes or hyperglycemia with order for basal insulin
Glucose Control: % patients with diabetes or hyperglycemia with orders for basal and nutritional insulin | up to 21 months
  Processes of care: % patients with diabetes or hyperglycemia with orders for basal and nutritional insulin
Nutrition: % patient-days without any diet order | up to 21 months
  Processes of care: % patient-days without any diet order
Nutrition: % pt-days NPO with insulin aspart ordered at same time | up to 21 months
  Processes of care:% pt-days NPO with insulin aspart ordered at same time
Venous thromboembolism (VTE): % pt-days with appropriate prophylaxis ordered based on risk and contraindications | up to 21 months
  Processes of care: % patient-days with appropriate prophylaxis ordered based on risk and contraindications
Venous thromboembolism (VTE):% pt-days with appropriate prophylaxis administered based on risk and contraindications | up to 21 months
  Processes of care: % pt-days with appropriate prophylaxis administered based on risk and contraindications
Venous thromboembolism (VTE): % ordered pharmacologic prophylaxis doses administered | up to 21 months
  Processes of care: % ordered pharmacologic prophylaxis doses administered
Pain Control: % pt-days with MED > 100 mg | up to 21 months
  Processes of care: % pt-days with MED > 100 mg
Pain Control: % patient-days with opioids ordered and no adjunctive medications ordered | up to 21 months
  Processes of care: % patient-days with opioids ordered and no adjunctive medications ordered
Pain Control:% pt-days with opioids administered and no Richmond Agitation-Sedation Scale (RASS) score recorded | up to 21 months
  Processes of care: % pt-days with opioids administered and no Richmond Agitation-Sedation Scale (RASS) score recorded
Antibiotic Management: % patient-days with patients on broad-spectrum gram-positive and broad-spectrum gram-negative antibiotics for > 72 hours | up to 21 months
  Processes of care: % pt-days with patients on broad-spectrum gram-positive and broad-spectrum gram-negative antibiotics for > 72 hours
Antibiotic Management: % pt-days with pts on broad-spectrum antibiotics for > 72 hours | up to 21 months
  Processes of care: % patient-days with patients on broad-spectrum antibiotics for > 72 hours
Delirium Management: % patient-days Confusion Assessment Method (CAM) positive | up to 21 months
  Processes of care: % patient-days Confusion Assessment Method (CAM) positive
Delirium Management: % patient-days of patients at high risk for delirium on sedatives | up to 21 months
  Processes of care: % patient-days of patients at high risk for delirium on sedatives
Delirium Management: % patient-days of patients at high risk for delirium on ramelteon | up to 21 months
  Processes of care: % patient-days of patients at high risk for delirium on ramelteon
Delirium Management: % patient-days of patients with hyperactive delirium on neuroleptics | up to 21 months
  Processes of care: % patient-days of patients with hyperactive delirium on neuroleptics
Vascular Access: % patient-days with central line in place | up to 21 months
  Processes of care: % patient-days with central line in place
Foley Care: % patient-days with Foley catheter in place | up to 21 months
  Processes of care: % patient-days with Foley catheter in place
Foley Care: % patient-days with Foley documented but not ordered | up to 21 months
  Processes of care: % patient-days with Foley documented but not ordered
Foley Care: % patient-days with Foley documented but Nurse Driven Protocol (NDP) not ordered | up to 21 months
  Processes of care: % patient-days with Foley documented but NDP not ordered
Telemetry: % patient-days of high risk patients without any telemetry | up to 21 months
  Processes of care: % patient-days of high risk patients without any telemetry bottom page 5 mock tables
Telemetry: % patient-days of low risk patients on telemetry > 72h | up to 21 months
  Processes of care: % patient-days of low risk patients on telemetry > 72h
Bowel Regimen: % pt-days of patients on opioids and no bowel regimen ordered | up to 21 months
  Processes of care: % pt-days of patients on opioids and no bowel regimen ordered
Bowel Regimen:% patient-days where on opioids, no bowel movement 2 or more days, and no bowel regimen administered | up to 21 months
  Processes of care: % patient-days where on opioids, no bowel movement 2 or more days, and no bowel regimen administered
Fall / Mobility: Patient Falls based on safety reports per 1000 patient-days | up to 21 months
  Safety Outcomes: Patient Falls based on safety reports per 1000 patient-days
Fall / Mobility: Falls with injury based on safety reports per 1000 patient-days | up to 21 months
  Safety Outcomes: Falls with injury based on safety reports per 1000 patient-days
Glucose Control: Patient-day-weighted mean glucose | up to 21 months
  Safety Outcomes: Patient-day-weighted mean glucose
Glucose Control: Proportion of glucose readings 70-180 mg/dL, mean per patient | up to 21 months
  Safety Outcomes: Proportion of glucose readings 70-180 mg/dL, mean per patient
Glucose Control: Proportion of patient-days with hypoglycemia | up to 21 months
  Safety Outcomes: Proportion of patient-days with hypoglycemia
Glucose Control: Proportion of patient-days with severe hypoglycemia | up to 21 months
  Safety Outcomes: Proportion of patient-days with severe hypoglycemia
Venous Thromboembolism: proportion of hospitalizations with hospital-acquired VTE | up to 21 months
  Safety Outcomes: proportion of hospitalizations with hospital-acquired VTE
Venous Thromboembolism: proportion of hospitalizations with VTE within 30 days of discharge | up to 21 months
  Safety Outcomes: proportion of hospitalizations with VTE within 30 days of discharge
Pain Control: proportion of hospitalizations with opioid induced depression of consciousness or respiration | up to 21 months
  Safety Outcomes: proportion of hospitalizations with opioid induced depression of consciousness or respiration
Pain Control: proportion of hospitalizations of patients on opioids who required narcan | up to 21 months
  Safety Outcomes: proportion of hospitalizations of patients on opioids who required narcan
Pain Control: proportion of hospitalizations with severe opioid-related adverse drug event | up to 21 months
  Safety Outcomes: proportion of patients on opioids who had rapid response, code blue, ICU transfer, Bipap, mechanical ventilation
Pain Control: proportion of hospitalizations of patients on opioids with any opioid-related Adverse Drug Event | up to 21 months
  Safety Outcomes: proportion of hospitalizations of patients on opioids with any opioid-related Adverse Drug Event
Pressure Ulcers: proportion of hospitalizations with hospital-acquired pressure ulcer | up to 21 months
  Safety outcomes: proportion of hospitalizations with hospital-acquired pressure ulcer
Pressure Ulcers: proportion of hospitalizations with pressure ulcer worsening in stage from admission to discharge | up to 21 months
  Safety outcomes: proportion of hospitalizations with hospital-acquired pressure ulcer worsening in stage from admission to discharge
Delirium Management: proportion of hospitalizations requiring mechanical restraints | up to 21 months
  Safety outcomes: proportion of hospitalizations requiring mechanical restraints
Delirium Management: proportion of hospitalizations requiring code gray and requiring security | up to 21 months
  Safety outcomes: proportion of hospitalizations requiring code gray and requiring security
Vascular Access: Central Line Associated Blood Stream Infection (CLABSI) per 1000 patient-days | up to 21 months
  Safety outcomes: Central Line Associated Blood Stream Infection (CLABSI) per 1000 patient-days
Foley Care: Central Line Associate Urinary Tract Infection per 1000 patient-days | up to 21 months
  Safety outcomes: Central Line Associate Urinary Tract Infection per 1000 patient-days
Telemetry: proportion of hospitalizations for rapid response for arrhythmia | up to 21 months
  Safety outcomes: proportion of hospitalizations for rapid response for arrhythmia

OTHER OUTCOMES:
Provider perceptions of safety, communication based on Agency for Healthcare Research and Quality (AHRQ) patient safety climate survey | up to 21 months
  perceived teamwork climate on hospital care units based on Agency for Healthcare Research and Quality (AHRQ) patient safety climate survey
Patient activation, engagement, satisfaction based on Patient Activation Measure (PAM 13) | up to 21 months
  Patient and caregiver perceptions of how well clinical team kept them safe based on Patient Activation Measure (PAM 13)
Usability of tools/ technology based on Health iTues survey | up to 21 months
  usability of technology- ease of use based on Health iTues survey
Effects on workflow | up to 21 months
  cognitive burden based on direct observations
Adherence to PSLL patient safety information technology tools | up to 21 months
  use of tool by providers and patients
Health care utilization | up to 21 months
  Length of stay of patients
Patient Reported Safety Concerns- MySafeCare reporting tool | up to 21 months
  Rate of submissions into the MySafeCare reporting tool per 1000 patient days (confidence interval)
Proportion of hospitalizations with code blue or rapid response | up to 21 months
  Other Clinical Outcomes: Proportion of hospitalizations with cardio-respiratory code or rapid response
Proportion of hospitalizations with ICU transfer | up to 21 months
  Other Clinical Outcomes: Proportion of hospitalizations with ICU transfer
Average time of discharge | up to 21 months
  time of discharge averaged
Patient Activation Measure (PAM-13) | up to 21 months
  Patient Activation as measured by the PAM 13 survey
30-day non-elective readmission | up to 21 months
  30-day non-elective readmission
Patient Satisfaction (HCAHPS) | up to 21 months
  Patient Satisfaction as measured by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS)

CONTACTS AND LOCATIONS:
Overall Officials: David W Bates, MD MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dykes PC, Burns Z, Adelman J, Benneyan J, Bogaisky M, Carter E, Ergai A, Lindros ME, Lipsitz SR, Scanlan M, Shaykevich S, Bates DW. Evaluation of a Patient-Centered Fall-Prevention Tool Kit to Reduce Falls and Injuries: A Nonrandomized Controlled Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2025889. doi: 10.1001/jamanetworkopen.2020.25889. PMID 33201236